CLINICAL TRIAL: NCT07257367
Title: Accuracy and Safety Assessment of Pressure Sensing Sheath Blood Pressure Monitoring Compared to Traditional Invasive and Non-invasive Blood Pressure Monitoring in Interventional Procedures: A Prospective, Single-Center, Self-Controlled Randomized Study
Brief Title: Pressure Sensing Sheath Blood Pressure Monitoring Compared to Traditional Methods in Interventional Procedures
Status: Recruiting | Type: Observational
Sponsor: Shanghai Fourth People's Hospital Tongji University (Other)
Responsible Party: Principal Investigator, Yibin Fang, MD, PhD, Shanghai Fourth People's Hospital Tongji University
Other Study IDs: ENDO TSP-BP; 2025110-002 (Other: Shanghai Fourth People's Hospital Ethics Committee); ENDO TSP-BP (Other: Shanghai Fourth People's Hospital)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure Monitoring; Neuroendovascular Procedures
Keywords: Pressure sensing sheath; Blood pressure monitoring; Invasive blood pressure; Neuroendovascular intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All enrolled patients will receive simultaneous blood pressure monitoring using both methods: (1) Pressure sensing sheath monitoring system inserted via radial artery, and (2) Traditional radial arterial line monitoring on the contralateral side combined with standard non-invasive blood pressure cuff monitoring. This is a self-controlled study design where each patient serves as their own control.
  Interventions: Device: Pressure Sensing Sheath Monitoring; Device: Radial Arterial Line Monitoring

INTERVENTIONS:
Device: Pressure Sensing Sheath Monitoring — Continuous invasive blood pressure monitoring via pressure sensing sheath inserted through radial artery during interventional procedure. The pressure sensing sheath integrates a miniature pressure sensor within the vascular access sheath, enabling simultaneous vascular access and continuous blood pressure monitoring.
Device: Radial Arterial Line Monitoring — Traditional invasive blood pressure monitoring via radial arterial catheterization (RAC) on the contralateral radial artery, combined with standard non-invasive blood pressure cuff monitoring. This serves as the gold standard comparator for blood pressure measurement accuracy.

SUMMARY:
This observational study aims to evaluate the accuracy and safety of pressure sensing sheath blood pressure monitoring compared to traditional invasive and non-invasive blood pressure monitoring methods during neuroendovascular interventional procedures.

The study will enroll 50 adult patients undergoing elective neuroendovascular procedures requiring general anesthesia and continuous invasive blood pressure monitoring. Blood pressure will be simultaneously measured using three methods: (1) pressure sensing sheath, (2) radial arterial line, and (3) non-invasive cuff monitoring.

The primary outcome is the accuracy of blood pressure measurements from the pressure sensing sheath compared to radial arterial line measurements. Secondary outcomes include the incidence of access site complications, procedure duration, patient comfort scores, and cost-effectiveness analysis.

This prospective, single-center study will be conducted at Shanghai Fourth People's Hospital Affiliated to Tongji University from August 2025 to May 2027.

DETAILED DESCRIPTION:
* Detailed Description for ClinicalTrials.gov Registration

  * BACKGROUND

    * Current State of Blood Pressure Monitoring in Interventional Procedures

Real-time, accurate hemodynamic monitoring is crucial during various interventional procedures. Currently, the clinical "gold standard" for continuous invasive arterial blood pressure monitoring is achieved through peripheral arterial catheterization (typically radial artery) connected to a pressure transducer, known as Radial Artery Catheterization (RAC). Although RAC provides beat-to-beat blood pressure data, it has several inherent limitations.

First, RAC insertion is an additional invasive procedure requiring extra time and technical skill, potentially delaying the start of the primary procedure. Studies have shown that RAC insertion requires an average of 10.7 minutes of additional time, with delays exceeding 80 minutes possible in complex cases. Second, the catheterization process may cause patient discomfort; research indicates that approximately 31.6% of patients experience pain after RAC insertion, with about 30% finding the pain bothersome. Additionally, RAC is associated with various potential complications, including radial artery occlusion (incidence approximately 5.5%), hand ischemia, infection, and thrombosis.

As an alternative, non-invasive blood pressure (NIBP) monitoring is widely used due to its convenience and safety. However, NIBP provides only intermittent readings and may fail to capture critical blood pressure fluctuations in rapidly changing hemodynamic scenarios. This is particularly important in neurointerventional procedures, where real-time blood pressure monitoring is essential for preventing and managing complications such as vasospasm and thrombosis.

### Pressure Sensing Sheath Technology

Given the limitations of traditional monitoring methods, pressure sensing sheath technology has emerged as an innovative blood pressure monitoring approach. This technology integrates a miniature pressure sensor within the vascular access sheath, enabling continuous invasive blood pressure monitoring while establishing vascular access. Theoretically, this approach can simultaneously address the time consumption, patient discomfort, and monitoring discontinuity associated with traditional methods.

Internationally, pressure sensing sheath technology, represented by EndoPhys Corporation, has received U.S. FDA 510(k) clearance and entered clinical use. Purdy et al. first published accuracy validation research on pressure sensing sheath technology in 2017. Froehler et al. completed the first prospective controlled trial (Clinical Trial Registration Number: NCT03239847) in 2018, initially confirming the clinical value of this technology in neurointerventional procedures. However, existing studies are primarily single-center, small-sample investigations focused mainly on European and American populations, with a lack of randomized controlled trial evidence.

### Study Rationale and Innovation

#### Filling Evidence Gaps

Currently, there is a lack of high-quality prospective randomized controlled trial evidence to systematically verify whether pressure sensing sheath monitoring is non-inferior to the gold standard RAC in accuracy, and to comprehensively compare safety, procedural efficiency, and patient-physician satisfaction. Existing international studies have relatively small sample sizes (20-40 cases), and their external validity and generalizability require further verification.

* Establishing Standards for Chinese Population

Vascular anatomical structures and hemodynamic characteristics show certain racial differences. Vascular diameter, elasticity, and blood pressure variability patterns in the Chinese population may differ from those in European and American populations. This study will be the first to systematically evaluate the accuracy and safety of pressure sensing sheath technology in a Chinese population, providing scientific evidence for establishing application standards and operational specifications suitable for Chinese clinical practice.

* STUDY OBJECTIVES

  * Primary Objective To assess the non-inferiority of the pressure sensing sheath blood pressure monitoring system compared to traditional radial arterial line invasive blood pressure monitoring combined with standard blood pressure cuff monitoring in terms of blood pressure reading accuracy during interventional procedures.
  * Secondary Objectives - To compare the safety of two monitoring methods

    - To evaluate procedural efficiency and operational convenience

    - To analyze patient comfort
* STUDY HYPOTHESIS

  * Primary Hypothesis The pressure sensing sheath monitoring system is non-inferior to traditional radial arterial line invasive blood pressure monitoring in measuring mean arterial pressure accuracy during interventional procedures, with the 95% limits of agreement between the two methods within the clinically acceptable range (±10 mmHg).
  * Secondary Hypothesis Pressure sensing sheath monitoring is superior to or equivalent to traditional radial arterial line monitoring in terms of safety, procedural efficiency, and patient comfort.
* STUDY DESIGN

This is a prospective, single-center, self-controlled randomized, non-inferiority clinical study.

The study will enroll patients undergoing elective transradial interventional procedures requiring continuous invasive blood pressure monitoring (meeting inclusion criteria without exclusion criteria). Using a self-controlled randomized design, each patient will simultaneously receive both pressure sensing sheath blood pressure monitoring (experimental group) and traditional radial arterial line invasive blood pressure monitoring combined with standard blood pressure cuff monitoring (control group). The primary study endpoint is at 7 days. By synchronously comparing the performance of both monitoring methods in the same patient, individual differences are eliminated, demonstrating that pressure sensing sheath monitoring is non-inferior to traditional radial arterial line invasive blood pressure monitoring systems, thereby providing a superior monitoring option for clinical practice.

### Randomization Scheme

Laterality Randomization: A random sequence will be generated to randomly determine whether the pressure sensing sheath monitoring system is inserted into the left or right radial artery, with the control group monitoring system inserted into the contralateral radial artery.

Monitoring Time Point Randomization: Block randomization design will be used to randomly determine specific blood pressure measurement time points within preset monitoring time windows, ensuring time synchronization and randomness of monitoring for both groups.

Experimental Group: Pressure sensing sheath monitoring system (inserted via radial artery)

Control Group: Traditional radial arterial line invasive blood pressure monitoring system combined with standard blood pressure cuff monitoring

---

## STUDY POPULATION

* Data Source This study's data will be collected from Shanghai Fourth People's Hospital Affiliated to Tongji University using a prospective, single-center data collection approach. Study subjects will be patients aged ≥18 years scheduled to undergo elective transradial interventional procedures requiring continuous invasive blood pressure monitoring according to standard medical operational procedures. Data collection period will be from September 15, 2025, to May 31, 2027, with an anticipated enrollment of 50 patients meeting inclusion criteria.
* Diagnostic Criteria

This study primarily targets patients requiring transradial interventional procedures with continuous invasive blood pressure monitoring. Disease diagnostic criteria include:

Indications for Interventional Procedures: According to relevant clinical guidelines and expert consensus, diseases requiring transradial interventional treatment primarily include acute cerebral infarction, aneurysms, arteriovenous malformations, carotid artery stenosis, and other cerebrovascular diseases. Specific diagnostic criteria reference the latest cerebrovascular disease diagnosis and treatment guidelines, including comprehensive evaluation of clinical symptoms, imaging examinations (CT/CTA/MRI/MRA/DSA), and laboratory test results.

Indications for Continuous Invasive Blood Pressure Monitoring: According to clinical needs and standard medical operational procedures, patients requiring radial arterial catheterization for invasive blood pressure monitoring include: interventional procedure patients requiring real-time, accurate blood pressure monitoring to guide treatment; patients with potentially unstable hemodynamics requiring close monitoring; patients requiring precise blood pressure control during procedures to prevent complications.

* Inclusion Criteria

  * Age ≥18 years
  * Patients scheduled for elective transradial interventional procedures requiring continuous invasive blood pressure monitoring
  * Patients who must undergo radial arterial catheterization for invasive blood pressure monitoring according to clinical needs and standard medical operational procedures
  * Patients who can understand the study purpose, voluntarily participate and sign informed consent, and are willing to undergo relevant examinations and clinical follow-up
* Exclusion Criteria

  * Patients with contraindications to radial artery access
  * Patients with hemodynamic instability
  * Patients requiring postoperative continuous invasive blood pressure monitoring
  * Patients unable to provide informed consent
  * Patients with known severe aortic or subclavian artery stenosis or occlusion
  * Patients with severe coagulation dysfunction (INR ≥2.0, platelet count <75×10⁹/L)
  * BMI >40 kg/m²
  * Severe heart failure (NYHA Class IV) or patients requiring emergency rescue with hemodynamic instability
* Withdrawal Criteria

  * Symptom deterioration or clinical complications preventing scheduled procedure
  * Subject wishes to pursue non-protocol treatment
  * Subject voluntarily withdraws from the study for any reason

    * STUDY ENDPOINTS
* Primary Endpoint

Mean Arterial Pressure (MAP) Agreement Analysis:

* Bland-Altman method to analyze agreement between pressure sensing sheath monitoring and radial artery monitoring
* Calculate 95% limits of agreement
* Evaluate mean and standard deviation of differences between the two methods
* Non-inferiority criterion: 95% limits of agreement within ±10 mmHg
* Synchronously evaluate agreement between pressure sensing sheath monitoring and standard blood pressure cuff monitoring as a reference comparison

  * Secondary Endpoints

Secondary Efficacy Endpoints:

1. Systolic (SYS) and Diastolic (DIA) Blood Pressure Agreement Analysis:

   - Separate Bland-Altman analysis for SYS and DIA
   * Calculate Pearson correlation coefficient and Lin's concordance correlation coefficient
   * Evaluate systematic bias and proportional bias
2. Blood Pressure Waveform Analysis:

   - Waveform morphology comparison (upstroke slope, downstroke characteristics, etc.)
   * Pulse pressure variability analysis
   * Waveform quality scoring (signal-to-noise ratio, artifact degree)
3. Procedural Efficiency Indicators:

   * Procedure preparation time: Time from patient entering operating room to start of radial artery puncture
   * Monitoring establishment time: Time from puncture initiation to obtaining stable blood pressure waveform
   * Impact on total procedure time

     * Safety Endpoints

Secondary Safety Endpoints:

1. Intraoperative Complications (intraoperative visit):

   * Puncture-related immediate complications: vasospasm or dissection, hematoma
   * Puncture failure rate
   * Significant hemodynamic changes
2. Postoperative Complications within 24 Hours:

   - Puncture site-related early complications: delayed bleeding, hematoma, vasospasm or dissection, vascular occlusion
   * Abnormal puncture site healing
   * Radial artery patency abnormalities (palpation, ultrasound)
3. Short-term Follow-up Complications (7 days post-procedure):

   - Puncture site delayed complications: infection, vascular occlusion, pseudoaneurysm
   * Persistent neurological impairment
   * Long-term radial artery patency (palpation, ultrasound)
4. Patient-Reported Outcome Measures:

   - Puncture site pain score (VAS 0-10 points)

   - Impact on daily activities

   ---

   ## STUDY PROCEDURES

   ### Visit Schedule

   The study consists of 4 visits: Visit 1 (enrollment visit), Visit 2 (intraoperative visit), Visit 3 (24 hours post-procedure), and Visit 4 (7 days post-procedure). All visits are clinical follow-ups.
   * Visit 1 (Enrollment Visit)

     - Informed consent

     - Demographic characteristics: name, gender, age, height, weight, body mass index, smoking history, drinking history, family history, hypertension, diabetes history, peripheral artery disease history, cerebrovascular disease history, coronary heart disease history, PCI history, dyslipidemia history, liver disease, kidney disease history, coagulation dysfunction history, neurological disease history, clinical manifestations (acute cerebral infarction, aneurysm, arteriovenous malformation, carotid artery stenosis, etc.)

     - Clinical indicators: blood pressure, heart rate, complete blood count, coagulation function, liver function, kidney function, electrolytes, blood glucose, electrocardiogram, cranial imaging (CT/CTA/MRI/MRA/DSA), carotid ultrasound, etc.

     - Concomitant treatments

     - Determine if inclusion criteria are met and if exclusion criteria exist; if patient qualifies, randomization will be performed and appropriate treatment strategy assigned
   * Visit 2 (Intraoperative Visit)

     - Patient symptoms

     - Concomitant treatments

     - Endpoint events and adverse events: puncture-related complications (vasospasm, hematoma formation, pseudoaneurysm, thrombosis, infection), blood pressure monitoring equipment failure, puncture failure, local pain, and others

     - Synchronous blood pressure monitoring data collection: MAP, SYS, DIA, and blood pressure waveform data from both pressure sensing sheath monitoring and traditional radial arterial line invasive blood pressure monitoring, as well as standard blood pressure cuff monitoring comparison data

     - Procedural efficiency indicators: procedure preparation time (time from patient entering operating room to main procedure start), total time required to establish stable invasive blood pressure monitoring, puncture success rate

     - Operator satisfaction score and patient comfort assessment
   * Visit 3 (24 Hours Post-Procedure) and Visit 4 (7 Days Post-Procedure)

     * Patient symptoms
     * Concomitant treatments
     * Endpoint events and adverse events: puncture site-related complications (delayed bleeding, hematoma, infection, vascular occlusion, pseudoaneurysm formation, neurological impairment), thrombotic events, and others
     * Safety assessment: puncture site healing status, radial artery patency examination (palpation, ultrasound), signs of local infection, neurological function assessment, patient-reported puncture site pain and discomfort scores (VAS score) (Visits 3 and 4)

       * DATA MANAGEMENT
   * Data Governance

   The study employs prospective data collection at 4 predetermined visit time points: Visit 1 (enrollment), Visit 2 (intraoperative), Visit 3 (24 hours post-procedure), and Visit 4 (7 days post-procedure). Standardized Case Report Form (CRF) templates ensure data collection consistency and completeness. Intraoperative blood pressure monitoring data will be synchronously collected to ensure temporal matching between pressure sensing sheath monitoring and traditional radial arterial line invasive blood pressure monitoring.

   ### Data Management Plan

   Detailed standard operating procedures for data collection will be established, clearly defining data collection content and requirements for each visit time point. For primary endpoint data, double data entry will be employed to ensure data accuracy. Data collection checklists will be established to ensure important data items are not missed. For blood pressure monitoring data, strict synchronous measurement standards will be established to ensure both monitoring methods are measured at the same time points under identical conditions.

   Multiple levels of data quality control measures will be implemented. Real-time data monitoring systems will validate and quality-check intraoperative blood pressure monitoring data. Data quality checkpoints will regularly verify completeness, accuracy, and consistency, with timely identification and correction of missing or abnormal data. Data anomaly identification and processing workflows will verify and correct abnormal data promptly. Source data verification mechanisms will ensure consistency between CRF data and source documents, guaranteeing data authenticity and traceability.

   ---

   ## BIAS CONSIDERATIONS

   This study fully considers various potential biases and control measures during design and implementation. To control information bias, the study employs standardized equipment calibration to reduce measurement errors, with all pressure monitoring equipment calibrated before use to ensure measurement accuracy, and standardized training to ensure data collection consistency. For selection bias, subjects are screened strictly according to inclusion and exclusion criteria to ensure study population homogeneity, with comprehensive follow-up plans to minimize loss to follow-up and detailed recording of reasons for incomplete visits.

   Confounding bias control is a key feature of this study, employing a self-controlled randomized design where each patient simultaneously receives both blood pressure monitoring strategies. By synchronously comparing the performance of both monitoring methods in the same patient, individual differences are effectively eliminated. Additionally, synchronous measurement of blood pressure data from both monitoring methods during the procedure eliminates the impact of temporal factors on results. To avoid outcome-driven bias, the study protocol predefines the primary endpoint analysis method as Bland-Altman agreement analysis, with non-inferiority criterion set as 95% limits of agreement within ±10 mmHg, avoiding post-hoc selection of the most favorable analysis method.

   ---

   ## STATISTICAL ANALYSIS PLAN

   ### Sample Size Estimation

   The target sample size for this study is 50 cases. This sample size was not determined through statistical calculation but was comprehensively considered based on relevant literature and study design characteristics. According to FDA guidance on medical device clinical trials, non-inferiority studies evaluating medical device accuracy can have relatively small sample sizes when using self-controlled designs.

   Referring to previous research on pressure sensing sheath technology, Purdy et al.'s 2017 accuracy validation study enrolled 20 patients, and Froehler et al.'s 2018 prospective controlled trial (Clinical Trial Registration Number: NCT03239847) enrolled 40 patients, both confirming the clinical value of this technology. Based on sample size requirements for Bland-Altman agreement analysis, relevant statistical literature recommends a minimum of 30-50 samples for methodological comparison studies to obtain reliable agreement assessment results.

   Since this study employs a self-controlled randomized design where each patient simultaneously receives both blood pressure monitoring strategies as their own control, individual variation is effectively eliminated, providing higher statistical power compared to traditional independent sample designs. Considering single-center study feasibility, expected study duration, and enrollment rate of interventional procedure patients, 50 cases can both meet statistical requirements and have good operability. This sample size references conventions from international similar medical device accuracy assessment studies and can provide sufficient evidence support for the primary study endpoint.

   ### Data Set Definitions

   According to study design and analysis objectives, the following data sets are defined:

   Efficacy Analysis Set: All subjects meeting inclusion criteria, without exclusion criteria, who complete synchronous intraoperative blood pressure monitoring. This data set is used for primary endpoint and secondary efficacy endpoint analysis.

   Safety Analysis Set: All subjects receiving at least one blood pressure monitoring method, used for safety endpoint analysis, including monitoring-related complication incidence and patient-reported puncture site pain and discomfort scores.

   If the target population for analysis is a subset of the data set, subsets will be marked as corresponding target populations for subgroup analysis based on different blood pressure ranges or procedure types.

   ### Missing Data Handling

   This study employs prospective design with strict visit arrangements and data quality control measures to minimize data missingness. Primary analysis uses complete case analysis, analyzing only subjects with complete paired blood pressure monitoring data to ensure synchronous measurement data completeness and comparability.

   For subjects with missed visits, investigators will record in detail reasons for incomplete visits and make efforts to obtain other relevant information from subjects. For lost-to-follow-up subjects, available clinical data or vital signs will continue to be collected from interventional centers, referring hospitals, general practitioners, etc., according to protocol. Lost-to-follow-up subjects will not be replaced. Sensitivity analysis will employ different missing data handling methods for comparison, including last observation carried forward, to evaluate the impact of missing data on study conclusions.

   ### Descriptive Analysis

   Comprehensive descriptive analysis will be performed on all collected variables to characterize main variable features. Continuous variables will be described using mean ± standard deviation or median (interquartile range) according to data distribution characteristics. Categorical variables will be described using frequencies and percentages.

   Baseline variable descriptive analysis includes subject demographic characteristics (name, gender, age, height, weight, body mass index), medical history (smoking history, drinking history, family history, hypertension, diabetes history, peripheral artery disease history, cerebrovascular disease history, coronary heart disease history, PCI history, dyslipidemia history, etc.), clinical indicators (blood pressure, heart rate, complete blood count, coagulation function, liver function, kidney function, electrolytes, blood glucose, electrocardiogram), imaging examination results, and concomitant treatment status. Endpoint variables including blood pressure monitoring data, procedural efficiency indicators, and safety events will also undergo corresponding descriptive analysis.

   ### Primary Analysis

   Hypotheses:

   - H0: The 95% limits of agreement for MAP differences between pressure sensing sheath monitoring and radial arterial line monitoring exceed ±10 mmHg

   - H1: The 95% limits of agreement for MAP differences between the two methods are within ±10 mmHg

   Primary analysis method employs Bland-Altman agreement analysis, calculating mean and standard deviation of differences between the two methods, creating Bland-Altman scatter plots, calculating 95% limits of agreement, and evaluating fixed and proportional bias. Non-inferiority judgment criterion is 95% limits of agreement within ±10 mmHg.

   Simultaneously, agreement evaluation will calculate Lin's concordance correlation coefficient and Pearson correlation coefficient, and create equivalence plots. As a reference comparison, agreement between pressure sensing sheath monitoring and standard blood pressure cuff monitoring will be synchronously evaluated. Since a self-controlled randomized design is employed where each patient serves as their own control, effectively eliminating inter-individual differences, primary analysis does not require adjustment for confounding factors.

   ### Sensitivity Analysis

   To evaluate study conclusion robustness, multiple sensitivity analyses will be performed, including:

   - Subgroup analysis of different blood pressure ranges, comparing pressure sensing sheath monitoring agreement performance in low, normal, and high blood pressure ranges

   - Comparative analysis of different data set definitions, comparing differences in results between efficacy analysis set and safety analysis set

   - Comparison of different missing data handling methods, evaluating result consistency between complete case analysis and other imputation methods

   - Agreement analysis stratified by measurement time points, evaluating the impact of temporal factors at different procedure stages on blood pressure monitoring agreement
   * Agreement analysis after excluding extreme values, evaluating the impact of outliers on primary conclusions

     * Safety Analysis

   Safety analysis will employ descriptive statistical methods, analyzed according to adverse event definitions and grading (NCI-CTCAE 4.0). Primary analysis focuses on monitoring-related complication incidence, including vasospasm, hematoma, infection, thrombosis, pseudoaneurysm, etc., as well as patient-reported puncture site pain and discomfort scores (VAS score).

   Complication incidence and severity will be analyzed by visit time point, including intraoperative complications (puncture-related immediate complications, puncture failure rate, significant hemodynamic changes), postoperative complications within 24 hours (delayed bleeding, hematoma, vasospasm or dissection, vascular occlusion, abnormal puncture site healing), and short-term follow-up complications (7 days post-procedure: infection, vascular occlusion, pseudoaneurysm, persistent neurological impairment).

   Safety event analysis will use frequencies and percentages for description. When necessary, Fisher's exact test or McNemar's test (for paired data) will be used to compare differences in monitoring method-related complication incidence.

   ---

   ## QUALITY CONTROL

   Quality control objectives for this study align with ICH guidelines, ensuring scientific validity, completeness, accuracy, and traceability of study data, with particular attention to quality control of blood pressure monitoring data precision and synchronization.

   ### Personnel Training

   All medical staff participating in the study will receive standardized training in pressure sensing sheath monitoring equipment operation to ensure operational consistency and accuracy. Training content includes: pressure sensing sheath monitoring system operational procedures, standard operations for traditional radial arterial line blood pressure monitoring, standardized data collection processes, adverse event identification and reporting, and study protocol requirements and procedures.

   Training will employ a combination of theoretical instruction and practical operation to ensure all research personnel proficiently master equipment operation skills, with effectiveness confirmed through assessment.

   ### Data Quality Control

   A comprehensive data quality control system will be established with regular data quality checks to ensure data completeness and accuracy. Real-time data monitoring will record and validate intraoperative blood pressure monitoring data in real-time, ensuring data collection accuracy and completeness. Data completeness checks will regularly verify completeness and logical consistency, promptly identifying and correcting missing or abnormal data. Data consistency verification will compare data consistency across different visit time points, ensuring data continuity and reliability. Key data validation will perform double verification of primary endpoint data, ensuring core data accuracy. Source data verification will ensure consistency between data and source documents, guaranteeing data authenticity and traceability.

   ### Equipment Calibration

   All pressure monitoring equipment must be calibrated before use to ensure measurement accuracy meets study requirements. Equipment standardization employs uniformly specified monitoring equipment to ensure consistent equipment performance. Regular calibration according to equipment manual requirements calibrates pressure transducers regularly, establishing equipment calibration archives. Calibration records detail each calibration time, results, and operator, ensuring calibration process traceability. Equipment maintenance ensures all monitoring equipment is in good working condition, with regular equipment maintenance and upkeep, and timely handling of equipment failures.

   ---

   ## ETHICS AND REGULATORY CONSIDERATIONS
   * Ethics Committee Review

   This protocol, written informed consent form, and materials directly related to subjects must be submitted to the Ethics Committee and receive written Ethics Committee approval before formally commencing the study. Investigators must submit continuing review reports one month before ethics approval letter expiration to apply for approval extension.

   Upon study suspension and/or completion, investigators must notify the Ethics Committee in writing. Investigators must promptly report all changes occurring in study work to the Ethics Committee (such as protocol and/or informed consent form amendments), and must not implement these changes without Ethics Committee approval, unless the changes are made to eliminate obvious and immediate risks to subjects. In such cases, the Ethics Committee will be notified.

   ### Informed Consent

   Investigators must provide subjects or their legal representatives with an easily understandable Ethics Committee-approved informed consent form and allow subjects or their legal representatives sufficient time to consider the study. Subjects may not be enrolled before obtaining signed written informed consent from subjects. During subject participation, subjects will be provided with all updated versions of informed consent forms and written information. Informed consent forms should be retained as important clinical trial documents for inspection.

   ### Confidentiality Measures

   Results from this project research may be published in medical journals, but personal information will be kept confidential according to legal and regulatory requirements. Unless required by relevant laws, patient personal information will not be disclosed. When necessary, government regulatory authorities, hospital ethics committees, and related personnel may inspect patient data according to regulations.

   ---
   * STUDY TIMELINE

   Study Period: September 15, 2025 to May 31, 2027

   Estimated Timeline:

   - Patient enrollment and data collection: September 2025 - December 2026
   * Data analysis and manuscript preparation: January 2027 - May 2027
   * Final report completion: May 2027

     * SIGNIFICANCE

   This will be the first prospective, self-controlled randomized trial in a Chinese population to systematically evaluate pressure sensing sheath blood pressure monitoring technology. Results will provide high-quality evidence for clinical application of this innovative monitoring technology, potentially improving blood pressure monitoring in interventional procedures, reducing patient discomfort and complications, and improving procedural efficiency. If non-inferiority is confirmed, this technology could become an important alternative for blood pressure monitoring in interventional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients scheduled for elective transradial interventional procedures requiring continuous invasive blood pressure monitoring
* Patients who must undergo radial arterial catheterization for invasive blood pressure monitoring according to clinical needs and standard medical operational procedures
* Patients who can understand the study purpose, voluntarily participate and sign informed consent, and are willing to undergo relevant examinations and clinical follow-up

Exclusion Criteria:

* Contraindications to radial artery access
* Hemodynamic instability
* Patients requiring postoperative continuous invasive blood pressure monitoring
* Failure to obtain informed consent
* Known severe aortic or subclavian artery stenosis or occlusion
* Severe coagulation dysfunction (INR ≥2.0, platelet count <75×10⁹/L)
* BMI >40 kg/m²
* Severe heart failure (NYHA Class IV) or patients requiring emergency rescue with hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing elective neuroendovascular interventional procedures requiring general anesthesia and continuous invasive blood pressure monitoring at Shanghai Fourth People's Hospital Affiliated to Tongji University. Target enrollment is 50 patients from September 2025 to December 2026.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Agreement of Mean Arterial Pressure Between Pressure Sensing Sheath and Radial Arterial Line | Intraoperative (duration of procedure, approximately 1-4 hours)
  Agreement analysis of mean arterial pressure (MAP) measurements between pressure sensing sheath monitoring and radial arterial line monitoring using Bland-Altman method. Non-inferiority criterion: 95% limits of agreement within ±10 mmHg. Synchronous comparison of both methods in the same patient to eliminate individual differences.

SECONDARY OUTCOMES:
Agreement of Systolic and Diastolic Blood Pressure | Intraoperative (duration of procedure, approximately 1-4 hours)
  Bland-Altman analysis of systolic (SBP) and diastolic (DBP) blood pressure agreement between the two monitoring methods. Calculate Pearson correlation coefficient and Lin's concordance correlation coefficient.
Procedural Efficiency | From patient entry to operating room until completion of procedure setup (approximately 10-30 minutes)
  Time required to establish stable blood pressure monitoring from puncture initiation, procedure preparation time, and impact on total procedure duration.
Incidence of Access Site Complications | From procedure start through 7 days post-procedure
  Composite of puncture-related complications including: vasospasm, hematoma, infection, thrombosis, pseudoaneurysm formation, vessel occlusion, and neurological impairment. Assessed at multiple time points: intraoperative, 24 hours post-procedure, and 7 days post-procedure.
Patient-Reported Puncture Site Pain Score | 24 hours and 7 days post-procedure
  Visual Analog Scale (VAS) pain score (0-10 points) for puncture site discomfort and impact on daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fourth People's Hospital Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Result] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Result] Rashid M, Kwok CS, Pancholy S, Chugh S, Kedev SA, Bernat I, Ratib K, Large A, Fraser D, Nolan J, Mamas MA. Radial Artery Occlusion After Transradial Interventions: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Jan 25;5(1):e002686. doi: 10.1161/JAHA.115.002686. PMID 26811162
- [Result] Froehler MT, Chitale R, Magarik JA, Fusco MR. Comparison of a pressure-sensing sheath and radial arterial line for intraoperative blood pressure monitoring in neurointerventional procedures. J Neurointerv Surg. 2018 Aug;10(8):784-787. doi: 10.1136/neurintsurg-2018-013769. Epub 2018 Feb 27. PMID 29487193
- [Result] Purdy PD, South C, Klucznik RP, Liu KC, Novakovic RL, Puri AS, Pride GL, Aagaard-Kienitz B, Ray A, Elliott AC. Use of a pressure sensing sheath: comparison with standard means of blood pressure monitoring in catheterization procedures. J Neurointerv Surg. 2017 Aug;9(8):766-771. doi: 10.1136/neurintsurg-2016-012536. Epub 2016 Jul 15. PMID 27422970